CLINICAL TRIAL: NCT03526003
Title: Effect of Position and Pneumoperitoneum on Respiratory Mechanics and Transpulmonary Pressure During Laparoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Amit Lehavi MD FANZCA, Director of Pediatric Anesthesia, Rambam Health Care Campus
Other Study IDs: 075-18
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Surgical patients: Adult patient scheduled for laparoscopic surgery under general anesthesia
  Interventions: Diagnostic Test: Measurement of esophageal pressure

INTERVENTIONS:
Diagnostic Test: Measurement of esophageal pressure — Measurement of esophageal pressure during posture changes and pneumoperotoneum

SUMMARY:
This study is an observational study measuring the esophageal pressure in anesthetized surgical patient undergoing changes in posture and pneumoperitoneum

DETAILED DESCRIPTION:
The study is a prospective observational study. Following approval by the Institutional Review Board, the study will be performed in a prospective, longitudinal cohort manner. Patients scheduled for elective laparoscopic surgery aged between 20 and 60 years will be included. Each participant signed an informed consent. Exclusion criteria included respiratory pathology, a body mass index lower than 18 or higher than 40 kg/m2, esophageal pathology and previous esophageal or pulmonary operation.

Following induction of anesthesia using fentanyl 2-5 microgram/kg, propofol 1-3 mg/kg and muscle relaxation with rocuronium 0.6-0.8 mg/kg, the trachea will be intubated using a 7-8 mm ID endotracheal tube. Mechanical ventilation in a volume controlled mode with a tidal volume 6-8 ml/kg and a PEEP of 5 cm of water will be initiated at a rate of 12-16 breaths per minute using an anesthesia machine (Fabius GS Premium, Drägerwerk AG & Co. KGaA, Lübeck, Germany). Balanced general anesthesia will be maintained by sevoflurane and fentanyl.

Esophageal balloon catheter will be placed according to manufacturer instructions 9. In brief, the stomach will be decompressed and suctioned with an 18 F orogastric tube. This tube will be also utilized to estimate the depth of the lower esophageal sphincter, a measure that will be corroborated with external simulation of the approximate distance from the gastric opening to the nares. A lubricated 86 cm long closed-tip catheter with a 9.5 cm long balloon catheter at its distal end will be gently inserted via one nostril and advanced into the esophagus. The calculated depth aiding in positioning the balloon at the lower third of the thoracic cavity at about 10 cm above the lower esophageal sphincter, as guided by catheter markings, will be the product of patient height x 0.288. This location had been verified by the external measurements at described above. An extension tubing will be attached to the Y piece at the proximal ending of the catheter and connected to a syringe and a pre-calibrated pressure transducer via a 3-way stopcock. One ml of air will be injected into the balloon so that it became semi inflated, and the tracing on the pressure monitor will be adjusted with additional small amounts of air until no flattening or damping will be noted in the pressure waveform. When properly positioned, the catheter will be secured with tape to prevent movement or extubation.

Esophageal pressure will be continuously measured via a calibrated pressure transducer system (Art-Line ,BioMetrix, Kiryat Mada, Jerusalem, Israel) connected to a patient monitor (Datex AS/3, Datex Ohmeda Medical Equipment, GE Healthcare, USA) and recorded using a designated computer software.

Esophageal pressure will be documented with the patient at horizontal position, and with the head up, operating table elevated 20 cm (anti Trendelenburg position) and head down, operating table lowill bed 20 cm (Trendelenburg position).

Following peritoneal access and trocar insertion, the peritoneal cavity will be gradually inflated with carbon dioxide by a laparoscopy insufflator (UHI-4 High Flow Insufflation Unit, Olympus Corporation Inc., Center Valley, PA, USA) and esophageal pressure will be recorded at a stable peritoneal pressure of 5, 10 and 15 mmHg. Following complete peritoneal inflation, the esophageal balloon catheter will be removed and recording terminated.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for laparoscopic surgery
* body mass index between 25 and 45

Exclusion Criteria:

* pregnancy
* contraindications for insertion of nasogastric tube

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective laparoscopic surgery aged between 20 and 80 years will be included. Each participant signed an informed consent. Exclusion criteria included respiratory pathology, a body mass index lower than 25 or higher than 45 kg/m2, esophageal pathology and previous esophageal or pulmonary operation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2019-05-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Changes in esophageal pressure | From immidiatly after induction of general anesthesia and mechanical ventilation to 10 minutes after initiation of pneumoperitoneum
  Effect of posture and pneumoperitoneum on esophageal pressure

IPD SHARING:
Plan to Share IPD: No
will not make ipd available

REFERENCES:
- [Background] Fish E, Novack V, Banner-Goodspeed VM, Sarge T, Loring S, Talmor D. The Esophageal Pressure-Guided Ventilation 2 (EPVent2) trial protocol: a multicentre, randomised clinical trial of mechanical ventilation guided by transpulmonary pressure. BMJ Open. 2014 Oct 6;4(9):e006356. doi: 10.1136/bmjopen-2014-006356. PMID 25287106
- [Background] Plataki M, Hubmayr RD. Should mechanical ventilation be guided by esophageal pressure measurements? Curr Opin Crit Care. 2011 Jun;17(3):275-80. doi: 10.1097/MCC.0b013e328344dda6. PMID 21326094